CLINICAL TRIAL: NCT05297721
Title: Determination of Nurses' Level of Knowledge on Skin Tears in Acute Care Hospitals: A Cross-Sectional Study
Brief Title: Nurses' Level of Knowledge on Skin Tears: A Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Hatice Yüceler Kaçmaz (Other)
Responsible Party: Sponsor-Investigator, Hatice Yüceler Kaçmaz, Principal Investigator, TC Erciyes University
Organization: TC Erciyes University (Other)
Other Study IDs: 328.IRB3.140
Record Dates: First submitted 2022-03-06; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Nurse's Role; Wound; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Wounds and Injuries; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurse: Nurses who (1) were employed as a nurse for at least 1 year, (2) cared for patients aged 65 and over and (3) agreed to participate in the study were included in the study.
  Interventions: Other: Knowledge

INTERVENTIONS:
Other: Knowledge — Measuring the level of knowledge about skin tears

SUMMARY:
Skin tears (ST) are one of the skin integrity problems encountered in healthcare settings with rates equal to or greater than pressure injuries. However, the importance of this problem has been emphasized in the literature in recent years. This study was conducted to determine the knowledge level of nurses about ST.

DETAILED DESCRIPTION:
The population of the study consisted of all nurses working in acute care hospitals in Turkey.

The sample size of the study was calculated as 384 nurses. The data of the study were collected in the form of online and paper-based surveys (an introductory information form and the Skin Tear Knowledge Assessment Instrumen)

ELIGIBILITY:
Inclusion Criteria:

* were employed as a nurse for at least 1 year
* cared for patients aged 65 and over
* agreed to participate in the study

Exclusion Criteria:

• nurses who filled in the data collection tools incompletely

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all nurses working in acute care hospitals in Turkey.
Sampling Method: Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Skin Tear Knowledge Assessment Instrument | one month
  Skin Tear Knowledge Assessment Instrument was developed by Van Tiggelen et al. (2021)

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided